CLINICAL TRIAL: NCT02666781
Title: The Contribution of Rostral Shift of Fluid to Postoperative Worsening of Obstructive Sleep Apnea Severity in Surgical Patients - A Prospective Cohort Study
Brief Title: Postoperative Rostral Fluid Shift and Obstructive Sleep Apnea
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Society of Anesthesia and Sleep Medicine (Unknown)
Responsible Party: Sponsor
Other Study IDs: 15-9507
Record Dates: First submitted 2016-01-11; First posted 2016-01-28 (Estimated); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Obstructive Sleep Apnea
Keywords: OSA, Surgery, Postoperative, Rostral Fluid Shift
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pilot Group: Postoperative surgical Patients with or without Obstructive Sleep Apnea
  Interventions: Other: ApneaLink Plus, BIA Device

INTERVENTIONS:
Other: ApneaLink Plus, BIA Device — The study is only observational. No interventions will be performed. ApneaLink Plus will be used to diagnose Obstructive Sleep Apnea in potential candidates and grade its severity on Postoperative night 2 in participants. A BIA Device will be used to detect segmental fluid shifts. A 3-D accelerometer will be used to detect head and neck position.

SUMMARY:
Patients with obstructive sleep apnea (OSA) are more likely to experience postoperative complications and impact significantly on healthcare resources. In the surgical population, the type and volume of IV fluid administration may contribute to the worsening of postoperative sleep apnea but the pathophysiological mechanisms have not been elucidated. Recent research from general population suggests that intravenous (IV) fluid administration worsens the severity of OSA by shifting of fluid from the legs to the neck thus increasing neck size and causing airway collapse. In this novel study, our objective is to examine the contribution of IV fluid administration and rostral fluid shift from the legs to the neck thereby leading to worsening of sleep apnea following surgery. In this prospective observational cohort study, 25 consecutive adult patients, requiring at least 2 days hospital stay, will be recruited. Following informed consent, patients will undergo portable home sleep study to determine the preoperative severity of sleep-disordered breathing. On the day of surgery, leg, neck and total body fluid volumes will be recorded, and patients will undergo general anesthetic. The results of this study will be used to design future clinical trials evaluating methods to decrease postoperative OSA worsening, as well as decreasing OSA-related postoperative complications.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common sleep-related breathing disorder, associated with increased morbidity and mortality. It is an independent risk-factor for post-operative cardio-respiratory complications and increased perioperative utilization of health care resources. In non-surgical patients, rostral fluid shift from the lower limbs to the neck has been identified as a pathophysiologic mechanism to explain OSA severity based on gender, increasing age, and in fluid-overload states. In this novel study, our objective is to examine the contribution of fluid shift from the lower limbs to the neck thereby leading to worsening of sleep apnea following surgery.

Objectives of the study

* Measure the change in the leg, neck and total fluid volume from preoperative baseline to the second postoperative day.
* Assess the impact of the change in neck fluid volume on neck circumference and postoperative AHI.

Similar to the patients with heart failure, renal failure and older men, we hypothesize the rostral shift of fluid from the lower limbs to the neck occurs in the postoperative period contributing to the postoperative worsening of OSA. In this study, we will perform serial measurements of segmental and total body water shifts occurring after surgery, at various time-points over two postoperative days. We will monitor indices such as the Apnea Hypopnea index (AHI) and oxygen desaturation index (ODI) to examine changes in the severity of OSA. Internal validity of our study will be made more robust by use of well-validated methods such as BIA for fluid measurements and portable PSG for OSA severity.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I to IV
* Undergoing elective non-cardiac surgery, requiring general anesthesia, lasting for 1-2 hours or more and requiring same day admission for a minimum of 2 days postoperatively.

Exclusion Criteria:

* Patients undergoing cardiac, intracranial surgery, procedures involving the neck such as cervical spine surgery, or carotid endarterectomy.
* Patients requiring epidural or spinal anesthesia for their surgery, as neuraxial blockade may impact fluid shifts from legs to neck and may confound our results.
* Prior history of vascular surgery in the lower limbs such as varicose vein surgery, vascular by-pass surgery or evidence of venous efficiency.
* Fluid overload states such as history of congestive heart failure, or renal failure will be excluded.
* Patients with metal implants in lower limbs or spine, due to possible interference with the leg impedance signals.
* Patients requiring urgent sleep physician referral (within four weeks) due to serious medical conditions or safety critical-occupations according to the 2011 Canadian Thoracic Society (CTS) guidelines e.g. unstable ischemic heart disease, recent cerebrovascular disease, congestive heart failure, obstructive/restrictive lung disease, pulmonary hypertension, hypercapnia respiratory failure.
* Pregnant or lactating patients, as the physiological mechanisms governing postoperative fluid shifts are different in this patient population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical patients attending the preoperative assessment clinic in Toronto Western Hospital (UHN) who will be undergoing elective non-cardiac surgery, requiring general anesthesia, lasting for 1-2 hours or more and requiring same day admission for a minimum of 2 days postoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-04-22 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2018-06-18 (Actual)

PRIMARY OUTCOMES:
Leg, neck and total body fluid volume on postoperative nights 1 and 2 | 48 hours
  Compartmental Fluids will be measured using an bioelectrical impedance device (BIA)

SECONDARY OUTCOMES:
Neck Circumference on Postoperative Nights 1 and 2 | 48 hours
  Neck circumference (in cm) will be assessed with a measuring tape and reported for correlation with other data
Apnea Hypopnea Index (AHI) on Postoperative Night 1 | 24 hours
  AHI will be measured as an indicator for the severity of Obstructive Sleep Apnea using an ApneaLink plus device.

CONTACTS AND LOCATIONS:
Overall Officials: Mandeep Singh, MD,FRCPC, Principal Investigator — Department of Anesthesia, Toronto Western Hospital- UHN, University of Toronto
Locations (1):
- Toronto Western Hospital- UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duran J, Esnaola S, Rubio R, Iztueta A. Obstructive sleep apnea-hypopnea and related clinical features in a population-based sample of subjects aged 30 to 70 yr. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):685-9. doi: 10.1164/ajrccm.163.3.2005065. PMID 11254524
- [Background] Mutter TC, Chateau D, Moffatt M, Ramsey C, Roos LL, Kryger M. A matched cohort study of postoperative outcomes in obstructive sleep apnea: could preoperative diagnosis and treatment prevent complications? Anesthesiology. 2014 Oct;121(4):707-18. doi: 10.1097/ALN.0000000000000407. PMID 25247853
- [Background] Chung F, Yegneswaran B, Liao P, Chung SA, Vairavanathan S, Islam S, Khajehdehi A, Shapiro CM. STOP questionnaire: a tool to screen patients for obstructive sleep apnea. Anesthesiology. 2008 May;108(5):812-21. doi: 10.1097/ALN.0b013e31816d83e4. PMID 18431116
- [Background] Ng SS, Chan TO, To KW, Ngai J, Tung A, Ko FW, Hui DS. Validation of a portable recording device (ApneaLink) for identifying patients with suspected obstructive sleep apnoea syndrome. Intern Med J. 2009 Nov;39(11):757-62. doi: 10.1111/j.1445-5994.2008.01827.x. Epub 2008 Nov 3. PMID 19220528
- [Derived] Lukachan GA, Chung F, Yadollahi A, Auckley D, Eissa M, Rahman N, McCluskey S, Singh M. Perioperative trends in neck and leg fluid volume in surgical patients: a prospective observational proof-of-concept study. Can J Anaesth. 2023 Feb;70(2):191-201. doi: 10.1007/s12630-022-02362-6. Epub 2022 Nov 30. PMID 36450944
- See also: Official Website for "STOP-Bang" Screening Questionnaire for Diagnosis of Obstructive Sleep Apnea — http://www.stopbang.ca